CLINICAL TRIAL: NCT06550557
Title: The Effect of a Counseling Intervention on Severe Nomophobia Among Health Care Providers: Randomized Controlled Clinical Trial
Brief Title: Counseling Intervention on Severe Nomophobia Among Health Care Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sarah Ahmed Abdelmoaty, assistant lecturer of family medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: nomophobia (MD-425-2022)
Record Dates: First submitted 2024-08-03; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Specific Phobia, Other
Keywords: nomophobia; health care providers; self-esteem; mental health
MeSH Terms: conditions — Phobia, Specific; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: pre intervention assessment of nomophobia score, mental health and self-esteem scores, then random allocation into intervention or control groups, intervention group received counselling sessions based on health belief model merged with smart phone action cues, post intervention scores were remeasured and compared to control group
Who Masked: Participant
Masking Description: participants into both the intervention and control groups didnot know of the other participants or the ongoing intervention nature
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- counseling group (Experimental): 1. assessement of nomophobia score, mental health and self-esteem scores.
  2. received 3 counselling sessions based on health belief model merged with smart phone action cues.
  3. assessment of nomophobia score, mental health and self-esteem scores post intervention
  Interventions: Behavioral: counselling sessions
- control group (No Intervention): assessment of nomophobia score, mental health and self-esteem scores at the same time interval of the intervention group, pre and post intervention

INTERVENTIONS:
Behavioral: counselling sessions — the counselling sessions were adopted from the health belief model with the cues of action depending on mobile phones as muting notifications, removing social media and using computers instead if possible.
  Arms: counseling group

SUMMARY:
Assess the effect of a counseling intervention adopted from heath belief model merged with multiple smart phone-based action cues on the level of nomophobia among participants with severe nomophobia Assess the effect of a counseling intervention adopted from heath belief model merged with multiple smart phone-based action cues on the level of nomophobia among participants with severe nomophobia

DETAILED DESCRIPTION:
In this study we seek to find if there is a relation between nomophobia level, self-esteem and mental health status, and discover whether a counseling intervention based on health belief model merged with smart phone-based action cues will decrease the level of nomophobia in participants with severe nomophobia.

through an intervention based on health belief model merged with multiple smart phone action cues employed on the intervention group during 3 counselling sessions

ELIGIBILITY:
Inclusion Criteria:

* Owning and actively using a smartphone.
* Understanding verbal English instructions.
* Willing to participate in a possible counseling session
* physicians currently working in kasr alainy hospital

Exclusion Criteria:

* Having any diagnosed psychiatric disorder.
* Participants taking medications that could affect psychological status e.g: B blockers, mood stabilizers.

Ages: 24 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-01-28 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Study the effect of the counseling program on severe nomophobia score among participants in the intervention group. | 18 months
  apply the counseling program and reassess the nomophobia level post-intervention by using the nomophobia questionnaire developed by Yildirim & Correia (2015). With a total of twenty statements on the questionnaire, responses were recorded on a 7-point Likert scale, with 7 representing strongly agree and 1 representing strongly disagree. The lack of nomophobia corresponded to a score of 20. Mild nomophobia was indicated by questionnaire scores ranging from 21 ≤ to < 60. On the other hand, scores between 60 and less than 100 suggested a moderate level of nomophobia, while scores between 100 and 140 indicated a severe level of nomophobia
Compare the level of nomophobia between intervention and control group post intervention. | 24 months
  apply the counseling program and comparing the nomophobia score with the control group post intervention at same time frame, by using the nomophobia questionnaire developed by (Yildirim & Correia, 2015) where severe nomophobes are those with a score above 100, comparing the post counseling sessions score between the intervention or the control group whether there was a significant decline in the nomophobia score.

SECONDARY OUTCOMES:
correlation between nomophobia scores, self-esteem scores and mental health scores | 18 months
  pre and post intervention nomophobia scores using the nomophobia questionnaire were correlated to the self-esteem scores using state self esteem questionnaire with r value expressed to show whether the correlation is positive or negative and it's strength.
  as well the nomophobia scores using nomophobia questionnaire were correlated to the mental health scores using the mental health inventory questionnaire, where positive r indicates positive correlation and negative r indicates an inverse correlation, the strength of the correlation is determined by the value of r.

CONTACTS AND LOCATIONS:
Overall Officials: sarah A Abdelmoaty, master, Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olson JA, Sandra DA, Chmoulevitch D, Raz A, Veissiere SPL. A Nudge-Based Intervention to Reduce Problematic Smartphone Use: Randomised Controlled Trial. Int J Ment Health Addict. 2022 May 17:1-23. doi: 10.1007/s11469-022-00826-w. Online ahead of print. PMID 35600564
- [Background] Notara V, Vagka E, Gnardellis C, Lagiou A. The Emerging Phenomenon of Nomophobia in Young Adults: A Systematic Review Study. Addict Health. 2021 Apr;13(2):120-136. doi: 10.22122/ahj.v13i2.309. PMID 34703533
- [Background] Wang Y, Wu AMS, Lau JTF. The health belief model and number of peers with internet addiction as inter-related factors of Internet addiction among secondary school students in Hong Kong. BMC Public Health. 2016 Mar 16;16:272. doi: 10.1186/s12889-016-2947-7. PMID 26983882